CLINICAL TRIAL: NCT02105363
Title: How Much Can the Thoracic and Lumbar Skin Slide? Unrecognized Cause of Epidural Catheter Placement Failure
Brief Title: How Much Can the Thoracic and Lumbar Skin Slide?
Status: Terminated | Type: Observational
Why Stopped: loss of research support
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Enrique Pantin, Professor, Department of Anesthesiology, Rutgers, The State University of New Jersey
Other Study IDs: 2013003345
Record Dates: First submitted 2014-02-25; First posted 2014-04-07 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Movement of Thoracic and Lumbar Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (20):
- Age 11-15
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 16-20
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 21-25
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 26-30
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 31-35
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 36-40
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 41-45
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 46-50
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 51-55
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 56-60
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- age 61-65
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 66-70
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 71-75
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 76-80
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 81-85
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 86-90
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 91-95
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 96-100
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 0-5
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back
- Age 6-10
  Interventions: Other: measure of skin movement on surface of the back; Other: Measurement of skin movement on surface of back

INTERVENTIONS:
Other: measure of skin movement on surface of the back
Other: Measurement of skin movement on surface of back

SUMMARY:
The investigators want to determine how much the skin on the back can move left to right of the midline and also up and down, in subjects presenting for procedure or in healthy volunteers. The investigators will do measurements on the back using samples of individuals in all age groups.

It is hypothesized that an explanation to late epidural failure could be related to excess back motion in individual subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Children age 0-17 and Adults 18 and older may participate
2. You agree to participate and sign the informed consent document

Exclusion Criteria:

1. Any type of back deformity
2. Tumor on back
3. Skin Disease on the back
4. Any condition that prevents skin measurements such as scleroderma

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals age 0-100
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Lumbar skin move greater than 4 cm laterally or cephala-caudal | Data entered day subject participates

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Pantin, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School; Ann Marie Lozano, RN, MSN, Study Chair — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Robert Wood Johnson Universtiy Hospital, New Brunswick, New Jersey, United States